CLINICAL TRIAL: NCT05651880
Title: Efficacy and Tolerance of Baricitinib, a JAK Inhibitor, in the Treatment of Refractory Non-infectious Non-anterior Uveitis
Acronym: JAKUVEITE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0420/HP
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Active Non-anterior Non-infectious Uveitis
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treated with baricitinib (Experimental): Patient treated with baricitinib at a dose of 4 mg per day, taken orally in the morning, with one tablet per day for 6 months.
  Interventions: Drug: Baricitinib 4 MG

INTERVENTIONS:
Drug: Baricitinib 4 MG — 4 mg per day for 6 months (For patients with creatinine clearance between 30 and 60 mL/min at baseline or during the study, the dosage of baricitinib will be 2 mg daily)

SUMMARY:
The aim of the study is to evaluate the efficacy of Baricitinib, a JAK1 and 2 inhibitor, in the management of non-infectious non-anterior uveitis refractory to at least one line of biotherapy (anti-TNF alpha, tocilizumab) after 6 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of non-anterior non-infectious uveitis, refractory to at least one line of biotherapy (anti-TNF alpha, tocilizumab)
* Need to stop biotherapy (anti-TNF alpha or tocilizumab) and conventional immunosuppressive drugs (mycofenolate mofetil, methotrexate, azathioprine, cyclosporine, interferon alpha 2a) for at least 10 days prior to the inclusion date

Exclusion Criteria:

* 1. Isolated anterior uveitis. 2. Infectious uveitis. 3. Severe uveitis threatening the visual prognosis and requiring emergency treatment with intravenous corticosteroids.

  4. Initial visual acuity > 1.3 LogMAR in at least one eye. 5. Corneal or lens opacity that prevents fundus visualization or may require cataract surgery during the study.

  6. Contraindication to baricitinib (OLUMIANT 2 and 4 mg film-coated tablets) : Hypersensitivity to the active substance or to any of the excipients.

  7. Contraindication to mydriasis. 8. Refractory glaucoma in either eye. 9. Monophthalmic patient. 10. Previous treatment with JAK inhibitors. 11. Intraocular corticosteroid injection (subconjunctival or laterobulbar) within 1 month prior to inclusion or intravitreal corticosteroid implant within 3 months prior to inclusion.

  12. Need for treatment with a biotherapy (anti-IL6, anti-IL6 receptor, anti-IL1, anti-IL12/IL23 anti-IL17, anti-BAFF) for extra-ocular involvement, during the entire study period.

  13. Treatment with OAT3 inhibitors with high inhibitory potential such as probenecid, leflunomide, teriflunomide 14. 14. Vaccination with a live or live attenuated vaccine within 15 days prior to inclusion 15. History of cancer within the previous 5 years, except non-metastatic squamous cell and basal cell carcinoma of the skin.

  16. Personal history of venous thromboembolic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete remission | 6 months

SECONDARY OUTCOMES:
Number of patients with complete remission | 1 month
Number of patients with complete remission | 3 months
Number of serious events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde LECLERCQ, MD, Principal Investigator — University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No